CLINICAL TRIAL: NCT05005039
Title: Bone Marrow Fat and Bariatric Surgery-Mediated Bone Loss
Acronym: ADIMOS-OB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0045; 2021-A01440-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-08-11; First posted 2021-08-13 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Bariatric Surgery in Postmenopausal Women

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese postmenopausal women who will undergo RYGB
- Obese postmenopausal women who will undergo SG

SUMMARY:
Results are inconsistent and further studies are needed to better understand the impact of bariatric surgery on the bone-BMA relationship depending on the type of bariatric surgery: RYGB vs. SG. Future studies are also needed to define the molecular mediators of bone loss and BMA changes. Several molecular mediators have been considered including gut hormones, adipokines, gonadal hormones and more recently G-CSF. However, the evidence to support any of these alone or in combination as primary mechanisms of bone loss is scant.

The study will be to explore potential changes in BMA after bariatric surgery and search for possible associated factors. Specifically, we want to investigate if such changes in BMFF differed in participants among different surgical types (RYGB vs. SG) and diabetic status. Secondly, we want to explore factors associated with BMFF changes including metabolic homeostasis (glycemic control and blood lipid levels), adipokines (leptin and adiponectin), calciotropic hormones (Ca++, PTH…), body composition parameters and bone markers (cross-laps, P1NP and sclerostin). We hypothesize that the BMFF would particularly decrease after RYGB compared to SG and that participants with T2D would have a larger decrease in BMFF than participants without T2D.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women (defined as last menses >12 months)

* Obesity with a BMI ≥ 35 kg/m²,
* Patients with an indication for bariatric surgery with two surgical techniques, RYGB and SG, but who have never had a bariatric surgery procedure previously,
* Enrollment will be stratified for each surgical techniques, RYGB and SG, by preoperative diabetes status, defined by having HbA1c >6.5% or a prior physician's diagnosis of diabetes plus use of an antidiabetic medication.
* Patients who have signed the informed consent.

Exclusion Criteria:

* women who were pre- and perimenopausal and men in order to minimize sex hormone and BMA changes unrelated to the surgical procedure.
* women who used medications known to impact bone metabolism or BMA, including bisphosphonates, teriparatide, denosumab, hormone replacement therapy (HRT) and oral glucocorticoids (>5mg prednisone equivalent daily for>10 days in the last 3 months.
* Other exclusion criteria included prior bariatric surgery, estimated glomerular filtration rate <30 mL/min,
* any contraindication to magnetic resonance imagery (MRI).

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Sample population will be 40 postmenopausal women suffering from obesity.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Variation in bone marrow fat fraction (BMFF) in % | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julien PACCOU, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France